

## INFORMED CONSENT FORM

Document Code: EY. FR. 16

Revision Date:24.03.2023

.Revision No:03

Version No:01

Page No: 1 / 6

## PLEASE READ THIS DOCUMENT CAREFULLY

| Dear | |
|-------|------|
| D 041 | <br> |

You are invited to participate in a study titled "Effect of kinesiology tape on pain, posture, balance and respiration in ankylosing spondylitis: a randomized controlled trial," conducted at Bursa Yuksek Ihtisas Training and Research Hospital. Before deciding whether or not to participate in this research, you need to understand why and how the research will be conducted, as well as the potential benefits, risks, and discomforts that may affect volunteer participants. Therefore, reading and understanding this form is of great importance. Please take time to read the following information carefully. You may discuss this information with your family, relatives, and/or doctor, if you wish. If there is anything you do not understand or is unclear, or if you would like more information, please ask us. If you agree to participate, a copy of this form, completed and signed by you, your doctor, and an authorized institutional witness, will be given to you for your records.

Participation in this research is entirely voluntary. You have the right to not participate or to withdraw from the study at any time. The responsible investigator may also exclude you from the study if deemed necessary. There will be no penalty or loss of any benefits you are entitled to in case of non-participation, withdrawal, or exclusion from the study. Information obtained from this study will be used solely for research purposes, and your personal information will be kept strictly confidential.

Participation in this research is entirely voluntary. You have the right to not participate or to withdraw from the study at any time after participating. In either case, there will be no penalty or loss of any benefits you are entitled to.

Research Supervisor (Name-Surname-Title-Signature) Professor Meliha Kasapoğlu Aksoy

#### Research aim:

The aim of this study is to examine the effect of the home exercise program given to patients diagnosed with Ankylosing Spondylitis on respiratory functions, balance, and pain.

#### How the research will be conducted:

You are in the group that will receive **home exercises**. Surveys and examinations will be performed face-to-face at the beginning and end of the exercise to determine the severity of Ankylosing Spondylitis and the effect of exercise treatment. The survey and examination will

Study Title: Effect of kinesiology tape on pain, posture, balance and. respiration in ankylosing spondylitis: a

randomized controlled trial



## INFORMED CONSENT FORM

Document Code: EY. FR. 16

Revision Date:24.03.2023

.Revision No:03

Version No:01

Page No: 2 / 6

take approximately **30 minutes**. The exercise program will be planned as home exercises for **5 weeks, 5 days a week, 3 sets of 10 repetitions per day**, and you will be shown how to perform the exercises.

**Location of the Research:** Bursa Yüksek İhtisas Training and Research Hospital, Physical Medicine and Rehabilitation Clinic

## **Participating researchers:**

Professor Meliha Kasapoglu Aksoy Busra Gokgun M.D.

**Duration of the research: 1 Year** 

**Expected number of volunteers: 70** 

# Benefits of participating in the study:

To provide improvement in complaints of pain, restricted mobility, balance disorders, stooping (kyphosis), and difficulty breathing caused by Ankylosing Spondylitis.

## Risks of participating in the study:

These treatments are routinely applied in patients with Ankylosing Spondylitis for the complaints of pain, restricted mobility, balance disorders, stooping, and difficulty breathing. There is **no risk** for you.

I, ......................[volunteer's name, surname (in their own handwriting)], have read the above text. I fully understand the scope and purpose of the study I am asked to participate in, and my responsibilities as a volunteer. I had the opportunity to ask questions and discuss the study and received satisfactory answers. I was also verbally informed about the potential risks and benefits of the study. I understand that I can withdraw from this study at any time without having to give any reason, and that my current treatment will not be negatively affected if I withdraw. Bu koşullarda;

- 1) I consent to participate in the aforementioned research voluntarily, without any pressure or coercion (and I also consent to my child's/guardian's participation in this study).
- 2) I consent to the access of my personal information by the individuals/institutions/organizations specified in the legislation, if deemed necessary, and
- 3) I consent to the use of the information obtained in this study for scientific publication, archiving, and, if necessary, its transfer outside of our country.

Study Title: Effect of kinesiology tape on pain, posture, balance and. respiration in ankylosing spondylitis: a

randomized controlled trial



## INFORMED CONSENT FORM

Do age No: 3 / 6 ΕY

| cument Code:<br>7. FR. 16 | I Revision Date:24 03 2023 Revision No:03 Vers | | Version No:01 | Pá |
|---|---|---|---|---|
| • | m | | | |
| Guardian's o<br>Name-Surna<br>Signature:<br>Address:<br>Phone numb | r o<br>m | er guardianship or custody<br>custody's (Handwritten)<br>e:<br>r, fax number, if any:<br>th/year):// | | |
| Name-Surna<br>Signature: Po | m<br>os | | from beginning t | o end |
| Name-Surna<br>Signature: | m | the statements<br>e:<br>th/year):/ | | |

NOTE: A copy of this form will remain with the volunteer, and another copy will be placed in the patient's file. A copy of the consent form obtained from healthy volunteers without a patient file or protocol number must be kept by the responsible investigator.

# **Contact person:**

Busra Gokgun M.D. +905384690900

Study Title: Effect of kinesiology tape on pain, posture, balance and. respiration in ankylosing spondylitis: a

randomized controlled trial



## INFORMED CONSENT FORM

Document Code: EY. FR. 16

Revision Date:24.03.2023

.Revision No:03

Version No:01

Page No: 4 / 6

### PLEASE READ THIS DOCUMENT CAREFULLY

| Dear | |
|------|------|
| Deal | <br> |

You are invited to participate in a study titled "Effect of kinesiology tape on pain, posture, balance and respiration in ankylosing spondylitis: a randomized controlled trial," conducted at Bursa Yuksek Ihtisas Training and Research Hospital. Before deciding whether or not to participate in this research, you need to understand why and how the research will be conducted, as well as the potential benefits, risks, and discomforts that may affect volunteer participants. Therefore, reading and understanding this form is of great importance. Please take time to read the following information carefully. You may discuss this information with your family, relatives, and/or doctor, if you wish. If there is anything you do not understand or is unclear, or if you would like more information, please ask us. If you agree to participate, a copy of this form, completed and signed by you, your doctor, and an authorized institutional witness, will be given to you for your records.

Participation in this research is entirely voluntary. You have the right to not participate or to withdraw from the study at any time. The responsible investigator may also exclude you from the study if deemed necessary. There will be no penalty or loss of any benefits you are entitled to in case of non-participation, withdrawal, or exclusion from the study. Information obtained from this study will be used solely for research purposes, and your personal information will be kept strictly confidential.

Participation in this research is entirely voluntary. You have the right to not participate or to withdraw from the study at any time after participating. In either case, there will be no penalty or loss of any benefits you are entitled to.

Research Supervisor (Name-Surname-Title-Signature) Professor Meliha Kasapoğlu Aksoy

#### Research aim:

The aim of this study is to examine the effect of the home exercise program given to patients diagnosed with Ankylosing Spondylitis on respiratory functions, balance, and pain.

Study Title: Effect of kinesiology tape on pain, posture, balance and. respiration in ankylosing spondylitis: a

randomized controlled trial



#### INFORMED CONSENT FORM

Document Code: EY. FR. 16

Revision Date:24.03.2023

.Revision No:03

Version No:01

Page No: 5 / 6

### How the research will be conducted:

You are in the group that will receive home exercises and Kinesio Tape (elastic band). Surveys and examinations will be performed face-to-face at the beginning and end of the exercise and tape treatment to determine the severity of Ankylosing Spondylitis and the effect of the treatment. The survey and examination will take approximately 30 minutes. The exercise program will be planned as home exercises for 5 weeks, 5 days a week, 3 sets of 10 repetitions per day, and you will be shown how to apply them. Additionally, Kinesio Tape will be applied by your doctor once a week for 5 weeks. This tape will remain on your skin for 5 days. Afterward, you will need to remove the tape at home.

**Location of the research:** SBU Bursa Yüksek İhtisas Training and Research Hospital, Physical Medicine and Rehabilitation Clinic

## Participating researchers:

Professor Meliha Kasapoglu Aksoy Busra Gokgun M.D.

**Duration of the research: 1 Year** 

**Expected number of volunteers: 70** 

## Benefits of participating in the study:

To provide improvement in complaints of pain, restricted mobility, balance disorders, stooping (kyphosis), and difficulty breathing caused by Ankylosing Spondylitis.

# Risks of participating in the study:

These treatments are routinely applied in patients with Ankylosing Spondylitis for the complaints of pain, restricted mobility, balance disorders, stooping, and difficulty breathing. There is **no risk** for you.

| l, | .[volunteer's name, | surname (in their ow | n handwriting)], have |
|---|---|---|---|
| read the above text. I fully und | derstand the scope | and purpose of the | study I am asked to |
| participate in, and my respon | nsibilities as a vol | unteer. I had the | opportunity to ask |
| questions and discuss the | study and receive | ed satisfactory ar | nswers. I was also |
| verbally informed about the p | ootential risks and | benefits of the stud | <b>ly.</b> I understand that I |
| can withdraw from this study a | at any time without | having to give any | reason, and that my |
| current treatment will not be ne | gatively affected if I | withdraw. | |
| Bu koşullarda; | | | |

Study Title: Effect of kinesiology tape on pain, posture, balance and. respiration in ankylosing spondylitis: a

randomized controlled trial

# T.C. Sağlık Bakanlığı Türkiye Kamu Həslənderi Krurmu

## BURSA YUKSEK IHTISAS TRAINING AND RESEARCH HOSPITAL

## INFORMED CONSENT FORM

Document Code: EY. FR. 16

Revision Date:24.03.2023

.Revision No:03

Version No:01

Page No: 6 / 6

- 1) I consent to participate in the aforementioned research voluntarily, without any pressure or coercion (and I also consent to my child's/guardian's participation in this study).
- 2) I consent to the access of my personal information by the individuals/institutions/organizations specified in the legislation, if deemed necessary, and
- 3) I consent to the use of the information obtained in this study for scientific publication, archiving, and, if necessary, its transfer outside of our country.

| Volunteer's (Handwritten) Name-Surname: Signature: Address: (Phone number, fax number, if any): Date (day/month/year):/ |
|---|
| For those under guardianship or custody Guardian's or custody's (Handwritten) Name-Surname: Signature: Address: Phone number, fax number, if any: Date (day/month/year):// |
| Organization official witnessing the approval process from beginning to end Name-Surname: Signature: Position: Date (day/month/year):// |
| Person making the statements Name-Surname: Signature: Date (day/month/year):/ |

NOTE: A copy of this form will remain with the volunteer, and another copy will be placed in the patient's file. A copy of the consent form obtained from healthy volunteers without a patient file or protocol number must be kept by the responsible investigator.

### **Contact person:**

Busra Gokgun M.D. +905384690900

Study Title: Effect of kinesiology tape on pain, posture, balance and. respiration in ankylosing spondylitis: a

randomized controlled trial